CLINICAL TRIAL: NCT05158088
Title: Video Laryngoscope Versus a USB Borescope Aided Endotracheal Intubation in Adults With Anticipated Difficult Airway
Brief Title: Video Laryngoscope Versus USB Borescope in Difficult Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdelghany ali, Lecturer of anesthesia and surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: N-15-2021/MSc
Record Dates: First submitted 2021-08-22; First posted 2021-12-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Intubation; Difficult or Failed
Keywords: Airway; Intubation; Videolaryngoscope; Borescope

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Borescope group (Active Comparator): Using an Endotracheal tube mounted over Borescope with the aid of conventional laryngoscope for intubation
  Interventions: Device: Borescope
- Videolaryngoscope group (Active Comparator): Using videolaryngoscope for intubation
  Interventions: Device: Video laryngoscope

INTERVENTIONS:
Device: Borescope — Endotracheal intubation using borescope
  Arms: Borescope group
Device: Video laryngoscope — Endotracheal intubation using video laryngoscope
  Arms: Videolaryngoscope group

SUMMARY:
Video Laryngoscope Versus a USB Borescope Aided Endotracheal Intubation in Adults With Anticipated Difficult Airway

DETAILED DESCRIPTION:
For patients allocated to the USB-borescope technique, a proper size endotracheal tube will be placed over the USB-borescope (with an external diameter of 5.5 mm) which will be coated externally with water-soluble lubricant. The proper size laryngoscope blade will be inserted. The USB-borescope will be placed through the oral cavity and will be advanced while tracking it on a mobile phone, it will be advanced to the glottic opening. If needed, rotation of USB-borescope and/or external laryngeal manipulation will be used to align it with the vocal cord.

For patients allocated to the intubation over Video Laryngoscope technique, video laryngoscope (Insighters insight is3) proper size blade will be placed and introduction of the Video Laryngoscope till viewing the glottis opening then insertion of a proper sized endotracheal tube

ELIGIBILITY:
Inclusion Criteria:

* 1.American Society of Anesthesiologist ASA physical status I-II patients. 2.Both genders. 3.Age18-60 years old 4.BMI <35 5.patients with El-Ganzouri score more than or equal to 4

Exclusion Criteria:

* Presence of pulmonary diseases
* Uncontrolled hypertension
* Ischemic heart disease
* Cervical spine fracture
* Limited mouth opening
* known to have tumors or polyps in the upper airway
* History of difficult intubation or difficult bag-mask ventilation
* Patients with difficult bag-mask ventilation after induction of anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Time of intubation | 5 minutes
  in seconds

SECONDARY OUTCOMES:
Blood pressure before intubation, every 5 minutes after intubation till 15 minutes after intubation | 15 minutes
  Systolic, diastolic, and mean arterial blood pressures
Heart rate Heart rate | 15 minutes
  Heart rate before intubation, every 5 minutes after intubation till 15 minutes after intubation
The degree of view clarity | 1 minute
  Cormack-Lehane grading
Incidence of complications | 48 hours
  Incidence of complications as bleeding, failure
Number of trials for correct endotracheal intubation | 2 minutes
  Number of trial till successful intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Egypt